CLINICAL TRIAL: NCT07248540
Title: Evaluation of Intravenous Magnesium Administration in the Treatment of Dysmenorrhea
Brief Title: IV Magnesium in the Treatment of Acute Dysmenorrhea
Acronym: IVMAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, md, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOP-IVMAG-DYSMENORRHEA
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; Magnesium Therapy; Pain Management
MeSH Terms: conditions — Dysmenorrhea; Agnosia | interventions — Magnesium Sulfate; dexketoprofen trometamol

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, parallel assignment clinical trial where participants are allocated into two groups to receive different intravenous treatments: 2 ampoules of magnesium sulfate or intravenous dexketoprofen. Each treatment is administered over 15 minutes, and pain outcomes are compared between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate 2 Ampoules (Experimental): Participants receive 2 ampoules (8 ml total) of intravenous magnesium sulfate diluted in 100 ml normal saline, administered over 15 minutes.
  Interventions: Drug: Magnesium Sulfate (2 Ampoules)
- Intravenous Dexketoprofen (Active Comparator): Participants receive 50 mg of intravenous dexketoprofen diluted in 100 ml normal saline, administered over 15 minutes.
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Magnesium Sulfate (2 Ampoules) — Intravenous administration of 2 ampoules (8 ml total) of magnesium sulfate diluted in 100 ml normal saline, infused over 15 minutes.
  Arms: Magnesium Sulfate 2 Ampoules
Drug: Dexketoprofen — Intravenous administration of 50 mg dexketoprofen diluted in 100 ml normal saline, infused over 15 minutes.
  Arms: Intravenous Dexketoprofen

SUMMARY:
This prospective, randomized, double-blind clinical trial aims to evaluate the analgesic efficacy of intravenous magnesium sulfate in women presenting to the emergency department with acute dysmenorrhea. Participants will be randomized into two groups receiving either 2 ampoules of magnesium sulfate or intravenous dexketoprofen. Pain levels will be assessed using the Visual Analog Scale (VAS) before and after treatment.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind clinical trial is designed to evaluate the analgesic effectiveness of intravenous magnesium sulfate in women aged 18 to 35 years presenting to the emergency department with acute dysmenorrhea. Participants will be randomly assigned to one of two treatment groups: 2 ampoules of magnesium sulfate or intravenous dexketoprofen.

All medications will be diluted in 100 ml of normal saline and administered intravenously over 15 minutes. Pain intensity will be assessed using the Visual Analog Scale (VAS) before treatment and 1 hour after administration. Secondary outcomes include patient satisfaction, vital sign changes, and adverse effects.

The study aims to compare the analgesic efficacy and safety profile of intravenous magnesium sulfate with that of a standard nonsteroidal anti-inflammatory drug (dexketoprofen) in the management of acute dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 to 35 years

Presenting to the obstetrics and gynecology emergency department with a diagnosis of primary dysmenorrhea

Having regular menstrual cycles within the last 6 months

Having a Visual Analog Scale (VAS) pain score of ≥6 at emergency admission

Providing written informed consent for participation in the study

Exclusion Criteria:

Patients with secondary dysmenorrhea or underlying gynecological pathology

Pregnancy or breastfeeding

Use of analgesics or muscle relaxants within the last 3 days

Known allergy to magnesium sulfate or dexketoprofen trometamol

History of renal failure, cardiac arrhythmia, or serious systemic disease

Inability to assess pain due to mental disability or communication disorder

Failure to provide informed consent for participation in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by Visual Analog Scale (VAS) | Baseline and 1 hour after intravenous treatment
  Pain severity will be assessed using the 0-10 Visual Analog Scale (VAS) before treatment and 1 hour post-treatment. The study will evaluate and compare the analgesic effect of two different doses of intravenous magnesium sulfate (2 ampoules vs. 3 ampoules) and compare both to intravenous dexketoprofen in women presenting with acute dysmenorrhea.

CONTACTS AND LOCATIONS:
Overall Officials: havva betül bacak, md, Principal Investigator — SBÜ Gaziosmanpaşa Training and Research Hospital
Locations (1):
- SBÜ Gaziosmanpaşa Training and Research Hospital, Gaziosmanpaşa, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No